CLINICAL TRIAL: NCT00038857
Title: Megadose CD34 Selected Progenitor Cells for Transplantation in Patients With Advanced Hematological Malignant Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-220
Record Dates: First submitted 2002-06-05; First posted 2002-06-07 (Estimated); Results first posted 2012-08-07 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Leukemia; Lymphoma
Keywords: Acute Myelogenous Leukemia; Acute Lymphocytic Leukemia; Myelodysplastic Syndrome; Chronic Lymphocytic Leukemia; Leukemia; Lymphoma; Non Hodgkin's Lymphoma; T cell depletion; CD34 selected progenitors cell; GVHD
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — Melphalan; Thiotepa; fludarabine; fludarabine phosphate; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CD34 PBPC (Experimental): CD34 peripheral blood progenitor cell (PBPC) transplants in 3 groups: 1) HLA-matched Sibling Transplant Patients; 2) Unrelated Donor Transplant Patients; 3) Haplo Identical Transplant Patients. Preparative regimen is 140 mg/m^2 Melphalan on day -8, 10 mg/kg Thiotepa on day -7, 160 mg/m^2 Fludarabine over 4 days on days -6, -5, -4, -3 and 1.5 mg/kg of Rabbit ATG a day times 4 over 4 days on days -6, -5, -4, -3.
  Interventions: Procedure: Megadose of CD34 Selected Progenitor Cells; Drug: Melphalan; Drug: Thiotepa; Drug: Fludarabine; Drug: Rabbit ATG

INTERVENTIONS:
Procedure: Megadose of CD34 Selected Progenitor Cells — Haploidentical peripheral blood progenitor cell (PBPC) transplants on Day 0.
Drug: Melphalan — 140 mg/m^2 on day -8
  Other Names: Alkeran
Drug: Thiotepa — 10 mg/kg on day -7
Drug: Fludarabine — 160 mg/m^2 over 4 days on days -6, -5, -4, -3
  Other Names: Fludarabine Phosphate; Fludara
Drug: Rabbit ATG — 1.5 mg/kg of Rabbit ATG a day times 4 over 4 days on days -6, -5, -4, -3.
  Other Names: Rabbit antithymocyte globulin; ATG; rATG; Genzyme; Thymoglobulin

SUMMARY:
Donor:

This clinical study will evaluate the feasibility of a purified CD34 peripheral blood progenitor cell (PBPC) transplants in patients with hematological malignancies.

The primary objectives of the study are to evaluate the recipient obtaining donor derived neutrophil engraftment and the incidence of acute graft versus host disease [GvHD] (grade III-IV).

Secondary objectives include assessments of recipient having donor derived platelet engraftment, incidence of graft failure and chronic GvHD, overall and disease free survival, clinical safety and device performance of the CliniMACS CD34 selection device.

DETAILED DESCRIPTION:
Donor Description:

Before taking part in this study, donors will have an evaluation that is the standard for any bone marrow or blood stem cell donor. These include standard blood tests, an electrocardiogram (EKG), and a chest X-ray. Donors will also be given a general health questionnaire that is given to all blood donors in the United States. It should take no more than 10 minutes to complete the questionnaire.

Donors in this study will receive standard mobilization therapy with daily G-CSF every 12 hours. The Granulocyte colony-stimulating factor (G-CSF) will be given as an injection under the skin. The mobilization phase starts on the first day that donors receive G-CSF and continues until the final day of the stem cell collection process (leukapheresis).

Donors in this study will receive Neupogen (white blood cell growth factor) to stimulate the immature blood cells. They will receive two injections, twice a day for four days. On the fourth day, assuming they have enough immature white blood cells, researchers will start the stem cell collection process (leukapheresis).

The stem cell collection will go from 1 to 4 days until enough immature cells have been collected, but will not be done on any day the donor's platelet count falls below 75,000. The stem cell is called a CD34(+) cell. These cells will then be processed over a cell-processing machine to try to purify the immature fraction of cells and remove the T-lymphocytes that are part of the fatal graft versus host disease. The T-cell is called a CD3(+) cell.

Leukapheresis, with later CD34(+) cell selection, will start on the day when circulating CD34(+) count is at a high enough level. Leukapheresis will continue until the appropriate count is reached. If the CD3(+) count is too high, adjustments will be made.

For those donors who cannot reach the collection goal in one series of collection attempts, researchers will wait until the donor recovers from the first stem cell collection and try again. If the donor is unable to reach the collection goal again, another attempt will be made with a different donor.

The blood thinner used for the procedure will be acid citrate dextrose (ACD). Heparin may be substituted when clinically needed. No additional blood thinners or additives should be added beyond those normally used during leukapheresis. A unique identification and labeling system shall be used to track the leukapheresis product from collection to infusion.

Samples will be taken from each leukapheresis product pre- and post-selection for quality analysis.

This is an investigational study. No more than 90 donors will take part in this study. All will be enrolled at M. D. Anderson.

Recipient Description:

Before taking part in this study, recipients will have standard evaluations to determine the stage of their disease. These may include bone marrow aspirations and biopsies and if necessary, CT scans and chest x-rays. All recipients will go through cardiopulmonary evaluation.

The recipients will have an allogeneic bone marrow transplant with pre-treatment of thiotepa, fludarabine, melphalan, and antithymocyte globulin. This will be followed by infusion of the peripheral blood progenitor cells.

Recipients will have daily follow-up exams in the hospital. Recipients will be evaluated at least one to five times per week after they leave until Day 100. After that, they will have evaluations at least once every three months until about one year and then once every six months.

The CliniMACS device is being provided by used of an investigational device exemption for the FDA. Without the CliniMACS device, this procedure would not be possible.

This is an investigational study. A total of 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female recipients must have histopathologically confirmed diagnosis of hematological or lymphatic malignancy in one of the following categories:
2. Acute Leukemia: Recipients must have acute leukemia in second or greater remission in relapse, or primary refractory disease. Acute leukemia (in first remission with poor risk factors and molecular prognosis; acute myelogenous leukemia (AML) with -5, -7, t(6:9), +8, -11q23 and Acute lymphoblastic leukemia (ALL) with Phil+ t(9:22), t(4:11) and secondary remission inclusive).
3. Chronic myelogenous leukemia: Chronic Myeloid Leukemia (CML) in accelerated phase, blast crisis or second chronic phase.
4. Myelodysplastic syndrome (in high and intermediate risk categories) - marrow blast > 10% on differential.
5. Non-Hodgkin's lymphoma in relapse
6. Refractory chronic lymphoid leukemia (CLL) - refractory to fludarabine based regimen, unrelated donor and haploidentical only
7. The recipient must be <=60 years old at time of registration.
8. The recipient must have a related donor haploidentical for human leukocyte antigen (HLA), A, B, C, or DR loci. They may be partial matched on the other haplotype.
9. Recovery from prior therapy, chemotherapy, or radiotherapy, as defined by: Eastern Cooperative Oncology Group (ECOG) performance status equal or less than 2; have recovered from the toxicity of prior major chemotherapy at the start of the preparative regimen on this protocol
10. Adequate cardiac and pulmonary function (Left ventricular ejection fraction (LVEF) >45%, Carbon Monoxide Diffusing Capacity (DL CO)>50% corrected for hemoglobin)
11. Serum creatinine <1.5 mg/dL or creatinine clearance >50 ml/min for those above serum creatinine of 1.5; serum bilirubin <2.0 mg/dL; Aspartate transaminase (AST)/alanine aminotransferase (ALT) <2* Upper limits of normal (ULN) (unless secondary to disease)
12. Females of childbearing potential must have a negative serum or urine beta-HCG test within three weeks of registration. Patients will be informed of the risk of not receiving adequate contraception.
13. No prior cancer within five years with the exception of surgically cured non-melanoma skin cancer or in situ cancer of the cervix
14. The recipient and/or the recipient's legal guardian must have been informed of the investigational nature of this study and have signed a consent form which is in accordance with Federal guidelines and the guidelines of the participating institution.
15. Donor age must be 4-80 years and weight greater than 20 kg.
16. Medical history and physical examination confirm good health status as defined by institutional standards
17. Seronegative for HIV Ag, HIV 1+2 Ab, Human T Cell Leukemia Virus (HTLV) I/II Ab, HbsAg, HbcAb (IgM [combination screening test] and IgG), HCV, RPR for syphilis within 30 days of apheresis collection - If positive for Hepatitis B or C or syphilis, the recipient must be notified - the recipient may proceed if PI, recipient and donor agree and there is no substitute donor
18. HLA matching criteria
19. Female donors of child-bearing potential must have a negative serum or urine beta-HCG test within three weeks of mobilization
20. Capable of undergoing leukapheresis, have adequate venous access, and be willing to undergo insertion of a central catheter should leukapheresis via peripheral vein be inadequate
21. Agreeable to second donation of PBPC (or a bone marrow harvest) should the patient fail to demonstrate sustained engraftment following the transplant
22. The donor, or legal guardian greater than 18 years of age, must have been informed of the investigational nature of this study and have signed a consent form in accordance with Federal Guidelines and the guidelines of the participating institution. If the donor is less than 18 years of age, parent or legal guardian consent must be obtained.
23. The prospective donor will be screened for cytomegalovirus (CMV) seroreactivity and a seronegative donor will be utilized if available when the patient is seronegative.

Exclusion Criteria:

1. Participation in other clinical trials which involve investigational drugs or devices that might influence the endpoints of this study
2. Evidence of active hepatitis (B and/or C) or cirrhosis
3. Neither the recipient nor the donor may be HIV positive
4. Presence of any other active, uncontrolled bacterial, viral or fungal infection.
5. Uncontrolled central nervous system (CNS) involvement with tumor cells
6. Documented allergy to murine proteins or iron dextran
7. The recipient is a lactating female or, if of child-bearing potential, is unwilling to implement adequate birth control.
8. Severe end-organ dysfunctions, particularly neurologic deficits detectable by clinical examination or significant intellectual impairment in metabolic disorders
9. Evidence of active infection (including urinary tract infection, or upper respiratory tract infection) or hepatitis (on screening).
10. Medical or physical reason which makes the donor unlikely to tolerate or cooperate with growth factor therapy and leukapheresis.
11. Factors that place the donor at increased risk for complications from leukapheresis or G-CSF therapy such as pulmonary hypertension, coronary artery disease, peripheral vascular disease, cerebral vascular disease.
12. Lactating female or, if of child-bearing potential, is unwilling to implement adequate birth control.
13. Donors who are hepatitis positive, Human T-cell lymphotropic virus type I (HTLVI) positive need consent of Principal Investigator and determination that this is the best donor.

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2001-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Champlin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period:October 1, 2001 to November 1, 2008. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Of the 29 participants enrolled, one participant was excluded from the trial and did not receive any treatment.
Groups:
- CD34 PBPC: Melphalan 140 mg/m^2 given IV for one day. Thiotepa 10 mg/kg given IV for one day. Fludarabine 40 mg/m^2 given IV daily for four days. Rabbit ATG 1.5 mg/kg given IV daily for four days. Stem Cell Infusion of CD34+ Selected Cells given on Day 0.
Period: Overall Study
Arm/Group | CD34 PBPC
Started | 29
Completed | 28
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | CD34 PBPC
Number analyzed (Participants) | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 36 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Absolute Neutrophil Count Engraftment
Description: Absolute neutrophil engraftment defined as first of 3 consecutive days with Absolute neutrophil count (ANC) equal to or more than 0.5 * 10^9/L. Baseline to Day 30 post transplant.
Time Frame: Day 0 up to Day 30
Population: Analysis per protocol.
Measure: Number; unit: participant
Groups:
- Melphalan + Thiotepa + Fludarabine + Rabbit ATG + CD34 PBPC: Melphalan 140 mg/m^2 given for one day. Thiotepa 10 mg/kg given for one day. Fludarabine 40 mg/m^2 given daily for four days. Rabbit ATG 1.5 mg/kg given daily for four days. Infusion of CD34+ Selected Cells given on Day 0.
Arm/Group | Melphalan + Thiotepa + Fludarabine + Rabbit ATG + CD34 PBPC
Number analyzed (Participants) | 28
participant | 21

ADVERSE EVENTS:
Time Frame: 7 Years, 1 Month (October 1, 2001 to November 1, 2008)
Arm/Group | CD34 PBPC
Serious Adverse Events (participants affected / at risk) | 21/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD34 PBPC (N=28)
Graft Failure (General disorders) | 6 (6)
Infection (Infections and infestations) | 17 (17)
Left Ureteral Obstruction (Renal and urinary disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 2 (2)
Elevated alanine aminotransferase (ALT) (Hepatobiliary disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Fever (General disorders) | 9 (9)
Disease Relapse (General disorders) | 4 (4)
Graft vs Host Disease (General disorders) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 2 (2)
Death (General disorders) | 4 (4)
Cardiac Failure (Cardiac disorders) | 1 (1)
Thrombotic Microangiopathy (Blood and lymphatic system disorders) | 1 (1)
Diffuse Alveolar Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Encephalopathy (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD34 PBPC (N=28)
Low Platelets (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Fever (General disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 10 (10)
Mucositis (Gastrointestinal disorders) | 11 (11)
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 14 (14)
Elevated Creatinine (Renal and urinary disorders) | 2 (2)
BK Virus (Infections and infestations) | 3 (3)
Hemorrhagic Cystitis (Renal and urinary disorders) | 6 (6)
Elevated Alkaline Phosphatase (Hepatobiliary disorders) | 1 (1)
Elevated Alanine Aminotransferase (Hepatobiliary disorders) | 1 (1)
Elevated Bilirubin (Hepatobiliary disorders) | 2 (2)
Infecrtion (Infections and infestations) | 14 (14)
Neutropenic Fever (General disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Fluid Overload (General disorders) | 1 (1)
Graft versus Host Disease (General disorders) | 7 (7)
Diplopia (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No